CLINICAL TRIAL: NCT01000116
Title: Fibrin Glue Versus Tacked Fixation in Laparoscopic Groin Hernia Repair. A Randomized Double-blind Placebo-controlled Trial.
Brief Title: Fibrin Glue Versus Tacked Fixation in Groin Hernia Repair (TAPP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Mette Astrup Madsen, M.D., Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJ-138
Record Dates: First submitted 2009-10-16; First posted 2009-10-22 (Estimated); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Inguinal Hernia; Femoral Hernia
Keywords: Tapp; Early pain; well-being; Seroma; Haematoma; Fibrin glue; tacks
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral; Pain; Seroma; Hematoma | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrin glue (Active Comparator)
  Interventions: Procedure: Tacks
- Tacks (Active Comparator)
  Interventions: Procedure: Fibrin glue

INTERVENTIONS:
Procedure: Fibrin glue — Tissucol 2 ml
  Arms: Tacks
Procedure: Tacks — Protacks
  Arms: Fibrin glue

SUMMARY:
In this study the researchers want to compare fibrin glue versus tacked fixation in fixation of the mesh in laparoscopic groin hernia repair. The primary endpoints are early pain in the first 3 days postoperative days. Moreover, the researchers investigate general well-being, fatigue, seroma, haematoma, postoperative nausea and vomiting. Thirdly, they are investigating chronic pain and clinical recurrence.

ELIGIBILITY:
Inclusion Criteria:

* unilateral groin hernia
* planned laparoscopic inguinal or femoral herniorrhaphy
* ASA I-III
* fluent Danish

Exclusion Criteria:

* converting to open operation
* low compliance
* daily use of morphine or similar drugs daily in the last month
* complications to the operation

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Early pain after operation | 1 month

SECONDARY OUTCOMES:
haematoma in groin region | day 10
seroma in groin region | day 10
fatigue | 10 days
discomfort | 6 month
Postoperative nausea and vomiting (PONV) | 10 days
Use of Analgesics at PACU | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Mette A Tolver, M.D., Principal Investigator — University Hospital Koege; Thue Bisgaard, M.D. DMSc, Principal Investigator — University Hospital Koege; Poul Juul, M.D., Principal Investigator — Private Hospital Hamlet; Jacob Rosenberg, M.D. DMSc, Principal Investigator — Herlev Hospital
Locations (1):
- Private Hospital Hamlet, Søborg, Denmark

REFERENCES:
- [Derived] Tolver MA, Rosenberg J, Juul P, Bisgaard T. Randomized clinical trial of fibrin glue versus tacked fixation in laparoscopic groin hernia repair. Surg Endosc. 2013 Aug;27(8):2727-33. doi: 10.1007/s00464-012-2766-6. Epub 2013 Jan 26. PMID 23355162